CLINICAL TRIAL: NCT03862417
Title: The Adult Degenerative Scoliosis Exercise Trial (Pilot Study)
Acronym: ADSET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00086262
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Degenerative Scoliosis
Keywords: Scoliosis; Exercise; Pain; Posture; Quality of life; Disability
MeSH Terms: conditions — Scoliosis; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the observation (control) group or the Schroth exercise treatment group using REDCAP.
  All outcomes will be measured at baseline and at a 3-month follow-up. Longer term effects will be assessed 3 months after the exercise program.
  The control group will be under observation for 3 months. The Schroth group will participate in weekly supervised sessions and a daily home program for 3 months. After 3 months, controls will undergo the same exercise protocol. This will allow examining exercise effects using these patients as their own controls and improve willingness for randomization.
Who Masked: Outcomes Assessor
Masking Description: Baseline exams will occur before randomization. Participants and therapists will be reminded not to discuss their group allocation. Evaluators will be blinded to group allocation. The statistician will also complete analyses blinded to which group received therapy or when they did.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth exercise group (Experimental): Will attend 5 1-hr long individual sessions to learn Schroth exercises and the home program. A 30-min. daily home program of 3 to 4 exercises will be progressed by the certified Schroth therapist using an algorithm. Patients will attend weekly 1-hr long group therapist-led exercise classes for 3 months. At each group class, adequate exercise performance will be assessed using the checklist. An algorithm guides the prescription of exercises intensity and progression from static to dynamic depending on the participant's ability. Prescription begins with Sitting on a Ball. If performed adequately, a more challenging exercise is attempted. The 3 most challenging exercises performed adequately as per the checklist will be prescribed with a detailed handout.
  Interventions: Other: Schroth exercises
- Control group (No Intervention): Observation without treatment or with previously prescribed pain medication is the current standard for adults with degenerative scoliosis not planning surgery.

INTERVENTIONS:
Other: Schroth exercises — An exercise program begun individually and then continued in groups.
  Other Names: Schroth
  Arms: Schroth exercise group

SUMMARY:
Adult degenerative scoliosis is the most common spine deformity in adults. Patients present a lateral curvature of the spine and vertebra rotation. Curves meeting indications for treatment affect 24% of the aging adult population. Adult scoliosis causes pain, curve progression, and cosmetic deformity affecting quality of life and function. Pain affects 90% of patients with AS. Other than surgery for severe cases and pain medication, very little non-operative treatments have been investigated. Scoliosis-specific exercises have shown promise in a single study in adults and in an Alberta adolescent study.

The goal of this pilot randomized controlled trial on the effect of Schroth exercises in adults with degenerative scoliosis compared to observation is to determine the feasibility of conducting a larger study. This study will help plan and secure funding for a larger study by examining the ability to recruit enough eligible participants, whether patients can follow the prescribed program session attendance and complete the home exercises prescribed. The early estimate the effects of the exercises on pain, quality of life, disability, deformity and posture measurements will help determine the potential of this approach and the likely success of a larger RCT. This study addresses a need of adults with degenerative scoliosis who do not meet surgical indications but still experience pain and disability by exploring a promising exercise approach.

DETAILED DESCRIPTION:
1.1 Adult degenerative scoliosis. Scoliosis is a 3D spine deformity including frontal curves, vertebral rotations, and sagittal changes.1 A curve >10o after 18 years of age is called Adult Scoliosis (AS) and is the most common adult spinal deformity.2 Degenerative AS arises from asymmetric disc and facet degeneration or due to leg length discrepancy, hip pathology, and osteoporosis.3 Most AS curves are lumbar or thoracolumbar.4 The prevalence of degenerative AS is higher than adolescent scoliosis, but estimates range widely at 2.4% - 68%56. The prevalence of curves >20° is 24%.7

AS causes pain, curve progression, radiculopathy, or cosmetic deformity affecting quality of life and physical function8-10. Pain affects 90% of patients with AS9. Adults with degenerative scoliosis present more pain than with idiopathic scoliosis.3 Severe radiculopathy (47%), claudication (9%), weakness (8%), myelopathy, and bowel/bladder dysfunction(1%) are also more common in adults with scoliosis.11 Sagittal imbalance in AS is strongly correlated with disability and low quality of life.12 Curve progression is common in AS at 2-6o/yr.13 It is thus relevant to offer treatments to prevent curve progression and the signs and symptoms above.

1.2 What treatment is available? There is an important lack of evidence about non-operative treatments for AS despite the recommendation of non-operative treatments are the first line for treating AS.8,14,15 This suggestion arise mostly because of the high complications rates with surgery and poor bone quality8. However, exercise has generally not been offered in studies comparing non-operative to operative care.8,14,15 The main goal of rehabilitation in AS is to decrease pain, improve function and slow disease progression to avoid surgery.16,17 Our review on exercises for AS18 found only one study with high risk of bias showing that 20 weeks of scoliosis specific exercises compared to general physiotherapy led to significantly more improved pain (by 3.2/10 pts), SRS-22 quality of life (by 0.7/5 for function, 0.9 pain, 0.5 self-image, 0.7 mental health and 1.0 for satisfaction with care), and Oswestry disability (by 12%). Only adults with idiopathic scoliosis were included in this study19 and exercises have not yet been tested in adults with degenerative scoliosis.

1.3 Rationale for Schroth treatment: Our award winning work with adolescent idiopathic scoliosis suggests that pain, self-image and back muscle endurance improvements, as well as, reduced curve progression result from short exercise programs.20-22 Schroth is a 3D autocorrection exercise aiming to correct posture.23 Schroth exercises are not yet routinely used for adults in Edmonton, but surgeons and patients have expressed interest for evidence on exercise. Patients routinely seek treatment options for smaller curvatures and inquire about less invasive treatments than surgery.

1.4 Schroth treatment: Posture corrections are achieved with the use of pressure, mirror and therapist verbal and tactile feedback.24,25 Schroth exercises aim to improve the ability to maintain correct posture through endurance and strength training.22 Schroth exercises include de-rotation, side shifting, and stretching to establish vertebral alignment, torsion respiratory exercises, and strengthening for postural muscles.26

2. Specific Aims: To conduct a pilot study for an RCT on the effect of Schroth exercises in adults with degenerative scoliosis compared to observation. Specific goals of the pilot are to: 2.1) Determine the recruitment and eligibility rate of patients for the RCT; 2.2) Demonstrate the feasibility of the assessment and treatment protocol by showing a high percent compliance with program attendance and home exercises and low study dropout rate; and 2.3) Estimate the effect size and variability for all outcomes to determine the sample size for the proposed RCT.

3. Methods and Materials

3.1 Subjects: Adults over 50 years old with degenerative scoliosis (n=20) with pain (>2/10) will be recruited from referrals to Dr. Eric Huang and James Mahood and using community ads. Other inclusion criteria are: (1) curves 15°-45°. Curves over 50° are surgical candidates, and will be excluded. Patients who have had cortisone or anesthetic injections within the last 3 months, surgery or presenting contra-indications to exercises (fractures, cancer, severe cardio-vascular co-morbidities, or osteopenia) will be excluded.

3.2 Procedures: Patients will be invited to participate at the Drs' clinics. Participants will be randomized to the observation (control) group or the Schroth exercise treatment group using REDCAP. All outcomes will be measured at baseline and at a 3-month follow-up. Longer term effects will be assessed 3 months after the exercise program. The primary outcome is pain at 3 months controlling for medication use.27 Secondary outcomes include: spine curve angles, vertebral rotation, SRS-22 questionnaire (self-image, mental health, function, and pain and total scores), posture (Surface Topography), Global Rating of Change (GRC), Oswestry Disability index, and muscle endurance (Sorensen test). At baseline, a physical exam will ensure participants can exercise safely. The control group will be under observation for 3 months. The Schroth group will participate in weekly supervised sessions and a daily home program for 3 months. After 3 months, controls will undergo the same exercise protocol. This will allow examining exercise effects using these patients as their own controls and improve willingness for randomization.

3.3.1 Schroth exercises treatment: During the first 2 weeks, participants will attend 5 1-hr long individual sessions to learn Schroth exercises and the home program, and to confirm independent adequate performance with a checklist.28 A 30-min. daily home program of 3 to 4 exercises will be prescribed and progressed by the certified Schroth therapist throughout the project using an algorithm26. Compliance will be monitored weekly using a logbook. Patients will attend weekly 1-hr long group therapist-led exercise classes for 3 months. Classes increase compliance and sense of social support.29,30 At each group class, adequate exercise performance will be assessed using the checklist.28 An algorithm guides the prescription of exercises intensity and progression from static to dynamic depending on the participant's ability.28 Prescription begins with Sitting on a Ball. If performed adequately, a more challenging exercise is attempted. If performance is not adequate, an easier exercise is attempted. The 3 most challenging exercises performed adequately as per the checklist will be prescribed with a detailed handout.28

3.3.2 Control intervention: Observation without treatment or with previously prescribed pain medication is the current standard for adults with degenerative scoliosis not planning surgery.

3.4 Co-interventions, contamination monitoring: Pain medication use will be monitored by a single score using the validated Medication Quantification Scale.27 Participants will be asked to refrain from using co-interventions. Co-intervention use will be monitored as well as any contamination where controls may attempt Schroth treatment.

3.5 Assessment: Evaluators will be blinded to group allocation and patients reminded not to divulge.

3.5.1 Self-Report Questionnaires: Demographic/History- Socio-demographics, medical history, symptoms and modifying factors will be self-reported at baseline only to describe participants.

Numeric Pain Rating and diagram- (Primary outcome). A scale from 0 to 10 (worst imaginable pain) will assess current, best, worst pain intensity in the last 24 hours, with documented reliability and validity.31 A body pain diagram will categorize the location of symptoms with high reliability.32

The Scoliosis Research Society (SRS-22r) is a quality of life questionnaire with 22 questions assessing 5 domains: function, pain, self-image, mental health (5 questions each), and satisfaction (2 questions).33 Scores correspond to the average of the items. The SRS-22 has adequate test-retest reliability, and validity with good correlations with SF-36, SF-12, and Oswestry scores.34

The Oswestry disability questionnaire assesses back related disability (/100 important disability) using 10 questions. The Oswestry is recommended in the core set in spinal research and presents adequate reliability, validity and responsiveness.35,36

Global Rating of Change- A 15-point global rating scale,35,37 will only be used at each follow-up. The scale ranges from -7 (very great deal worse) to +7 (very great deal better).

3.5.2 Physical Exam: A physiotherapist blind to group assignment, will determine curve type28 and assess the range of motion for lower extremities, leg length (supine) and asymmetry in the forward bend test (with scoliometer).38,39 Lumbar and thoracic spinal range-of-motion will be recorded using double inclinometers: flexion, extension and side flexions. The Sorensen's test will assess back extensor endurance as the time the torso is maintained horizontal against gravity.40

3.5.3 3D ultrasound imaging- Standing 3D Ultrasound scans of the spine will be obtained without radiation exposure in a positioning frame. An experienced evaluator will extract curve angle, and apical vertebra rotations from de-identified images with high reliability and interchangeability with radiographs measurements has been shown.41-44

3.5.4 Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. ST parameters will be extracted in Matlab by digitizing 15 reference points on de-identified scans. The parameters quantifying the external trunk deformity are: cosmetic score composed of a weighted average of the shoulder angle, scapula angle and waist asymmetry, the trunk twist, and kyphotic and lumbar indices and angles from the sagittal view.45,46 We found parameters have adequate discriminative validity and sensitivity to change.47 Asymmetry maps will also be monitored.48-50

3.6. Analyses: Objective 1: Recruitment rates will be calculated as the percent of patients enrolled out of all patients invited. Eligibility rate corresponds to the percentage of patients meeting the selection criteria out of all patients assessed at clinics. Objective 2: Compliance will be calculated as the percentage of visits attended and percent prescribed home exercises reported performed. Drop-out rate will be calculated as the percentage of enrolled patients not completing the study. Objective 3: Cohen's D effect sizes and sample size needed will be estimated for all outcomes51,52 targeting a power of 0.80 with alpha of 0.05 using the observed change and variability from intention-to-treat analyses. Where available MCID will inform sample size estimation.

4. Significance: Adult degenerative scoliosis is a chronic and often painful condition, with a profound effect on patients.3,53 The Schroth exercise method is less invasive than current treatments (injections, surgery). Our review suggest that exercises can be effective to limit pain, disability and other deficits.18 RCTs on Schroth exercises for AS are needed. Clinicians and patients from the scoliosis clinic demand research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50 years old with degenerative scoliosis (n=20) with pain (>2/10). Other inclusion criteria are: (1) curves 15°-45°.

Exclusion Criteria:

* Curves over 50° are surgical candidates, and will be excluded. Patients who have had cortisone or anesthetic injections within the last 3 months, surgery or presenting contra-indications to exercises (fractures, cancer, severe cardio-vascular co-morbidities, or osteopenia) will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Percent of patients enrolled out of all patients invited.

SECONDARY OUTCOMES:
Eligibility rate | 1 year
  Percentage of patients meeting the selection criteria out of all patients assessed at clinics.
Compliance | 1 year
  Percentage of exercise visits attended
Adherence | 1 year
  Percent prescribed home exercises reported performed
Drop out rate | 1 year
  Percentage of enrolled patients not completing the study.

OTHER OUTCOMES:
Pain intensity assessed bhy the | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  A numeric pain rating scale from 0 to 10 (worst imaginable pain) will assess current, best, worst pain intensity in the last 24 hours, with documented reliability and validity.
Pain location | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  A body pain diagram will categorize the location of symptoms with high reliability
Scoliosis Research Society 22r scores | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Quality of life questionnaire with 22 questions assessing 5 domains: function, pain, self-image, mental health (5 questions each), and satisfaction (2 questions).33 Scores correspond to the average of the items. The SRS-22 has adequate test-retest reliability, and validity
Oswestry disability questionnaire | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  assesses back related disability (/100 important disability) using 10 questions. The Oswestry is recommended in the core set in spinal research and presents adequate reliability, validity and responsiveness.
15-point global rating scale, | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  A 15-point global rating scale, will only be used at each follow-up. The scale ranges from -7 (very great deal worse) to +7 (very great deal
Lumbar and thoracic spinal range-of-motion | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  will be recorded using double inclinometers: flexion, extension and side flexions
Sorensen test | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  The Sorensen's test will assess back extensor endurance as the time the torso is maintained horizontal against gravity.
Curve angle, and apical vertebra rotations | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Standing 3D Ultrasound scans of the spine will be obtained without radiation exposure in a positioning frame. The curve angle and rotation are extracted semi automatically by digitizing the location of the laminae on either side of the spine on each vertebra.
Cosmetic Score | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. ST parameters will be extracted in Matlab by digitizing 15 reference points on de-identified scans. One of the parameters quantifying the external trunk deformity is the cosmetic score composed of a weighted average of the shoulder angle, scapula angle and waist asymmetry, the trunk twist, and kyphotic and lumbar indices and angles from the sagittal view.45,46
Back surface rotation | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. Back surface rotation is obtained by dividing the full torso model in 90 cross-section and measuring the angle of the tangent to the most prominent points on the back surface of each cross-section. Back surface rotation corresponds to the range between the most rotated section to the left and to the right of the patient.
Centroid 3D deviations | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. Centroid deviation is obtained by dividing the full torso model in 90 cross-section and measuring the 3D coordinate of the centroid of each cross-section. The centroid deviation summary parameter corresponds to the distance between the largest deviations in 3D.
composite cosmetic Index (CCI) | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. The Waistline Height Index, Waistline Depth Index, Waistline Area Index, Waist Area Index, and hump index (α) are combined into a composite cosmetic Index (CCI) according to Qiu et al Spine 2010 35 (18) E882-8
Max deviation from asymmetry analysis | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. The ST scan of each full torso will be analyzed to calculate the best plane of symmetry by minimizing the distances between the torso and its reflection about the plane of symmetry. Distance between the torso and its reflection will measured and displayed as deviation color maps. The Root Mean Square of all deviations of the asymmetry maps for patches with deviations exceeding the 9.33mm threshold will be calculated. As per Ghaneei BMC Musculoskelet Disord. 2018 Oct 24;19(1):385.
RMS of the deviations from asymmetry analysis | 3 months, 6 months in Schroth group, 3 months, 6 months, 9 months in Control group
  Full-torso surface topography (ST) - Four Minolta 910 Laser Scanners and a positioning frame will be used to record full-torso ST scans. The operator will acquire scans blind to treatment groupings. The operator will position the subjects, mark reference points, and scan. The ST scan of each full torso will be analyzed to calculate the best plane of symmetry by minimizing the distances between the torso and its reflection about the plane of symmetry. Distance between the torso and its reflection will measured and displayed as deviation color maps. The Root Mean Square of all deviations of the asymmetry maps for patches with deviations exceeding the 9.33mm threshold will be calculated. As per Ghaneei BMC Musculoskelet Disord. 2018 Oct 24;19(1):385.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Parent, PT PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Faculty of Rehabilitation Medicine, Dept. Physical Therapy, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No